CLINICAL TRIAL: NCT01361152
Title: Long-Term Comparison of Fixed- and Mobile-Bearing Total Knee Arthroplasties in Patients With Osteoarthritis Younger Than Fifty Years of Age
Brief Title: Long-Term Comparison of Fixed- and Mobile-Bearing Total Knee Arthroplasties (TKAs) in Patients With OA ≤50 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor and Director, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fixed- and Mobile TKA
Record Dates: First submitted 2011-05-17; First posted 2011-05-26 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty; fixed-bearing; mobile-bearing; long-term
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed-bearing group (Experimental): Fixed-bearing group
  Interventions: Device: anatomic modular fixed-bearing
- Mobile-bearing group (Experimental): Mobile-bearing group
  Interventions: Device: low contact stress rotating platform mobile-bearing

INTERVENTIONS:
Device: anatomic modular fixed-bearing — anatomic modular (AMK; DePuy) fixed-bearing prosthesis
  Other Names: AMK
  Arms: Fixed-bearing group
Device: low contact stress rotating platform mobile-bearing — low contact stress rotating platform (LCS RP; DePuy) mobile-bearing prosthesis
  Other Names: LCS RP
  Arms: Mobile-bearing group

SUMMARY:
The purpose of the prospective study was to evaluate the minimum fifteen year follow-up of prospective total knee arthroplasties performed in patients younger than fifty years of age with osteoarthritis, using fixed- and mobile-bearing knee prostheses in the same patients, to compare

1. functional scores
2. rates of radiographic failure
3. revision rates
4. survivorship

DETAILED DESCRIPTION:
The randomized prospective comparison of fixed- and mobile-bearing total knee designs in the same patients younger than fifty years of age is limited. The purpose of this study was to compare the long-term clinical and radiographic results of fixed- and mobile-bearing total knee arthroplasties in patients younger than fifty years of age with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* End-stage osteoarthritis of the knee joint requiring total knee arthroplasty with bilateral disease

Exclusion Criteria:

* Inflammatory disease
* Patient with other Lower extremity disease which may affect functional outcome
* Neurologic disease effecting patients lower extremity
* Revision surgery
* Patient not medically cleared for bilateral surgery

Ages: 29 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 1993-04; Primary Completion 1996-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Knee Society Knee Score | 18 years
  change in knee score will be compared with initial score, until follow up of 18 years

SECONDARY OUTCOMES:
Improvement in the range of motion | 18 years
  change in the range of motion of knee joint will be compared with the initial value, until follow up of 18 years.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, MD, Study Director — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hosptial, Seoul, South Korea